CLINICAL TRIAL: NCT01876511
Title: Phase 2 Study of MK-3475 in Patients With Microsatellite Unstable (MSI) Tumors
Brief Title: Study of MK-3475 in Patients With Microsatellite Unstable (MSI) Tumors (Cohorts A, B and C)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J1365 (Cohort A, B and C); MK-3475-016 (Other: Merck); NA_00085756 (Other: JHMIRB)
Record Dates: First submitted 2013-06-10; First posted 2013-06-12 (Estimated); Results first posted 2020-01-07 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: MSI Positive Colorectal Cancer; MSI Negative Colorectal Cancer; MSI Positive Non-Colorectal Cancers
Keywords: microsatellite unstable (MSI); microsatellite stable (MSS); MLH 1; MSH 2; MSH 6; PMS2
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A: MSI Positive Colorectal Cancer (Experimental)
  Interventions: Drug: MK-3475
- Cohort B: MSI Negative Colorectal Cancer (Experimental)
  Interventions: Drug: MK-3475
- Cohort C: MSI Positive Non-Colorectal Cancer (Experimental)
  Interventions: Drug: MK-3475

INTERVENTIONS:
Drug: MK-3475 — MK-3475 10 mg/kg every 14 days

SUMMARY:
This study will be looking at whether MK-3475 (an antibody that blocks negative signals to T cells) is effective (anti-tumor activity) and safe in three different patient populations. These include: 1. patients with MSI positive colon cancer, 2. patients with MSI negative colon cancer and 3. patients with other MSI positive cancers.

ELIGIBILITY:
Inclusion Criteria:

* Cohort A only: Patients with microsatellite instability (MSI) positive colorectal cancer
* Cohort B only: Patients with MSI negative colorectal cancer
* Cohort C only: Patients with MSI positive non-colorectal cancer -
* Have measurable disease
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 1
* Adequate organ function as defined by study-specified laboratory tests
* Must use acceptable form of birth control through the study and for 28 days after final dose of study drug
* Signed informed consent form
* Willing and able to comply with study procedures
* Agree to have a biopsy of participants' cancer
* Patients with colon cancer must have received at least two prior cancer therapy regimens.
* Patients with other cancer types must have received at least one prior cancer therapy
* Progressive disease

Exclusion Criteria:

* Patients with uncontrolled intercurrent illness, including but not limited to ongoing or active infection, systematic congestive heart failure, unstable angina pectoris, cardiac arrhythmia or psychiatric condition that would limit compliance with study requirements.
* Patients who have had chemotherapy or biological cancer therapy within 2 weeks prior to the first dose of study drug
* Patients who have had radiation within 2 weeks prior to the first dose of study drug
* Patients who have undergone major surgery within 4 weeks of dosing of investigational agent
* Patients who have received another investigational product or investigational device within 4 weeks prior to receiving study drug
* Patients who have received any of the following concomitant therapy: Interleukin-2 (IL-2), interferon, or other non-study immunotherapy regimens, immunosuppressive agents, other investigational therapies or chronic use of systemic corticosteroids within one week prior to first dose of study drug
* Patients who have received a live vaccine within 4 weeks prior to or after any dose of MK-3475 (exception: inactivated flu vaccines)
* Patients who have received growth factors, including but not limited to granulocyte-colony stimulating factor (G-CSF), granulocyte macrophage-colony stimulating factor (GM-CSF), erythropoietin, etc. within 2 weeks of study drug administration
* Patient who have had prior treatment with anti-PD-1 (anti-programmed cell death protein 1), anti-PD-L1, anti-PD-L2, anti-CD137, anti-OX-40, anti-CD40, or anti-CTLA-4 antibodies
* Patients with history of any autoimmune disease:inflammatory bowel disease, (including ulcerative colitis and Crohn's Disease), rheumatoid arthritis, systemic progressive sclerosis (scleroderma), systemic lupus erythematosus (SLE) autoimmune vasculitis, central nervous system (CNS) or motor neuropathy considered to be of autoimmune origin.
* Patients who have known history of infection with HIV, hepatitis B, or hepatitis C
* Patients with evidence of interstitial lung disease
* Systemically active steroid use
* Patients on home oxygen
* Patients with oxygen saturation of <92% on room air by pulse oximetry
* Pregnant or lactating
* Conditions, including alcohol or drug dependence, or intercurrent illness that would affect the patient's ability to comply with study visits and procedures
* Patient with known active central nervous system metastases and/or carcinomatous meningitis.
* Patients with primary brain tumors.
* Requires any other form of systemic or localized antineoplastic therapy while on study
* Has any tissue or organ allograft
* Patients with history of allogeneic hematopoeitic stem cell transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dung Le, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (7):
- United States (7):
  - Stanford University, Stanford, California
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Investigator Thoracic and Gastrointestinal Oncology Branch, Center for Cancer Research, NIH, Bethesda, Maryland
  - Ohio State University, Columbus, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - University of Pennsylvania, Abramson Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Le DT, Durham JN, Smith KN, Wang H, Bartlett BR, Aulakh LK, Lu S, Kemberling H, Wilt C, Luber BS, Wong F, Azad NS, Rucki AA, Laheru D, Donehower R, Zaheer A, Fisher GA, Crocenzi TS, Lee JJ, Greten TF, Duffy AG, Ciombor KK, Eyring AD, Lam BH, Joe A, Kang SP, Holdhoff M, Danilova L, Cope L, Meyer C, Zhou S, Goldberg RM, Armstrong DK, Bever KM, Fader AN, Taube J, Housseau F, Spetzler D, Xiao N, Pardoll DM, Papadopoulos N, Kinzler KW, Eshleman JR, Vogelstein B, Anders RA, Diaz LA Jr. Mismatch repair deficiency predicts response of solid tumors to PD-1 blockade. Science. 2017 Jul 28;357(6349):409-413. doi: 10.1126/science.aan6733. Epub 2017 Jun 8. PMID 28596308
- [Background] Le DT, Uram JN, Wang H, Bartlett BR, Kemberling H, Eyring AD, Skora AD, Luber BS, Azad NS, Laheru D, Biedrzycki B, Donehower RC, Zaheer A, Fisher GA, Crocenzi TS, Lee JJ, Duffy SM, Goldberg RM, de la Chapelle A, Koshiji M, Bhaijee F, Huebner T, Hruban RH, Wood LD, Cuka N, Pardoll DM, Papadopoulos N, Kinzler KW, Zhou S, Cornish TC, Taube JM, Anders RA, Eshleman JR, Vogelstein B, Diaz LA Jr. PD-1 Blockade in Tumors with Mismatch-Repair Deficiency. N Engl J Med. 2015 Jun 25;372(26):2509-20. doi: 10.1056/NEJMoa1500596. Epub 2015 May 30. PMID 26028255

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort A: MSI Positive Colorectal Cancer | Cohort B: MSI Negative Colorectal Cancer | Cohort C: MSI Positive Non-Colorectal Cancer
Started | 41 | 25 | 47
Stages 1 and 2 | 24 | 25 | 21
Completed | 18 | 0 | 16
Not Completed | 23 | 25 | 31
Not completed — Disease Progression-clinical/radiologic | 11 | 24 | 16
Not completed — Death (unrelated) | 3 | 0 | 2
Not completed — Drug-related Toxicity | 5 | 1 | 6
Not completed — Patient Decision | 3 | 0 | 6
Not completed — Physician Decision | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: MSI Positive Colorectal Cancer | Cohort B: MSI Negative Colorectal Cancer | Cohort C: MSI Positive Non-Colorectal Cancer | Total
Number analyzed (Participants) | 41 | 25 | 47 | 113
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 31 | 15 | 30 | 76
  >=65 years | 10 | 10 | 17 | 37
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 9 | 23 | 51
  Male | 22 | 16 | 24 | 62
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2 | 4
  Not Hispanic or Latino | 39 | 25 | 44 | 108
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 1 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 3 | 1 | 7
  White | 34 | 21 | 44 | 99
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Immune-related Progression Free Survival (irPFS) at 20 Weeks in MSI Positive and Negative Colorectal Adenocarcinoma Participants Using Immune Related Response Criteria (irRC) During Stages 1 and 2
Description: For Cohorts A and B: irPFS rate is defined as the percentage of patients with disease progression (irPD or relapse from irCR as assessed using irRC criteria) or death due to any cause at 20 weeks. Per irRC criteria, Complete Response (irCR) is the disappearance of all target lesions, Partial Response (irPR) is a decrease in tumor burden by 50% or greater by a consecutive assessment at least 4 weeks after first documentation, Stable Disease (irSD) is the failure to meet criteria for irCR or irPR (in absence of irPD), Progressive Disease (irPD) is at least 25% increase in tumor burden relative to nadir. Estimation based on the Kaplan-Meier curve.
Time Frame: 20 weeks
Population: It was a pre-specified objective to complete this objective in Cohort A and B only. Per protocol during stages 1 and 2, the study enrollment goal was 25 for Cohort A and B. However, only 24 subjects were enrolled in Cohort A. Additional subjects for this study were enrolled during the second expansion portion of this protocol.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: MSI Positive Colorectal Cancer | Cohort B: MSI Negative Colorectal Cancer
Number analyzed (Participants) | 24 | 25
percentage of participants | 88 [75 to 100] | 12 [4 to 36]

2. Primary Outcome: Immune-related Objective Response Rate in MSI Positive and Negative Colorectal Adenocarcinoma Participants Using Immune Related Response Criteria (irRC) During Stages 1 and 2
Description: For Cohorts A and B: Immune-related Objective Response Rate (irORR) is defined as the percentage of patients achieving a complete response (irCR) or partial response (irPR) based on irRC criteria. Per irRC criteria, Complete Response (irCR) is the disappearance of all target lesions, Partial Response (irPR) is a decrease in tumor burden by 50% or greater by a consecutive assessment at least 4 weeks after first documentation.
Time Frame: 28 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: MSI Positive Colorectal Cancer | Cohort B: MSI Negative Colorectal Cancer
Number analyzed (Participants) | 24 | 25
percentage of participants | 67 [45 to 84] | 0 [0 to 14]

3. Primary Outcome: Immune-related Progression Free Survival (irPFS) at 20 Weeks in MSI Positive Non-colorectal Adenocarcinoma Participants Using Immune Related Response Criteria (irRC) During Stages 1 and 2
Description: For Cohort C: irPFS rate is defined as the percentage of patients with disease progression (irPD or relapse from irCR as assessed using irRC criteria) or death due to any cause at 20 weeks. Per irRC criteria, Complete Response (irCR) is the disappearance of all target lesions, Partial Response (irPR) is a decrease in tumor burden by 50% or greater by a consecutive assessment at least 4 weeks after first documentation, Stable Disease (irSD) is the failure to meet criteria for irCR or irPR (in absence of irPD), Progressive Disease (irPD) is at least 25% increase in tumor burden relative to nadir. Estimation based on the Kaplan-Meier curve.
Time Frame: 20 weeks
Population: It was a pre-specified objective to complete this objective in Cohort C only. Per protocol during stages 1 and 2, the study enrollment goal was 21 for Cohort C. Additional subjects for this study were enrolled during the second expansion portion of this protocol.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort C: MSI Positive Non-Colorectal Cancer
Number analyzed (Participants) | 21
percentage of participants | 67 [49 to 90]

4. Primary Outcome: Objective Response Rate in MSI Positive Solid Tumor Malignancies Using Response Evaluation Criteria in Solid Tumors (RECIST 1.1)
Description: For Cohorts A and C: Objective Response Rate (ORR) is defined as the percentage of patients achieving a complete response (CR) or partial response (PR) based on RECIST 1.1 criteria. CR = disappearance of all target lesions, PR is =>30% decrease in sum of diameters of target lesions.
Time Frame: 28 months
Population: It was a pre-specified objective to complete this objective in Cohort A and C only.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: MSI Positive Colorectal Cancer | Cohort C: MSI Positive Non-Colorectal Cancer
Number analyzed (Participants) | 41 | 47
percentage of participants | 54 [37 to 69] | 55 [40 to 70]

5. Primary Outcome: Progression Free Survival (PFS) at 20 Weeks in MSI Positive Solid Tumor Malignancies Using Response Evaluation Criteria in Solid Tumors (RECIST 1.1)
Description: For Cohorts A and C: PFS is defined as the percentage of patients with disease progression (PD or relapse from CR as assessed using RECIST 1.1 criteria) or death due to any cause at 20 weeks. Per RECIST 1.1 criteria, CR = disappearance of all target lesions, Partial Response (PR) is =>30% decrease in sum of diameters of target lesions, Progressive Disease (PD) is >20% increase in sum of diameters of target lesions, Stable Disease (SD) is <30% decrease or <20% increase in sum of diameters of target lesions. Estimation based on the Kaplan-Meier curve.
Time Frame: 20 weeks
Population: It was a pre-specified objective to complete this objective in Cohort A and C only.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: MSI Positive Colorectal Cancer | Cohort C: MSI Positive Non-Colorectal Cancer
Number analyzed (Participants) | 41 | 47
percentage of participants | 75 [63 to 90] | 68 [56 to 83]

6. Secondary Outcome: Overall Survival (OS)
Description: OS will be measured from date of first dose until death or end of follow-up (OS will be censored on the date the subject was last known to be alive for subjects without documentation of death at the time of analysis). Estimation based on the Kaplan-Meier curve.
Time Frame: 4 years
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Cohort A: MSI Positive Colorectal Cancer | Cohort B: MSI Negative Colorectal Cancer | Cohort C: MSI Positive Non-Colorectal Cancer
Number analyzed (Participants) | 41 | 25 | 47
Weeks | NA [151.86 to NA] — NA means that the median overall survival and upper bound confidence interval was not reached. | 36.71 [21.29 to 69.43] | 148.86 [94.71 to NA] — NA means that the upper bound confidence interval was not reached.

7. Secondary Outcome: Immune-related Progression Free Survival (irPFS) at 28 Weeks in MSI Positive and Negative Solid Tumor Malignancies Using Immune Related Response Criteria (irRC)
Description: irPFS rate is defined as the percentage of patients with disease progression (irPD or relapse from irCR as assessed using irRC criteria) or death due to any cause at 28 weeks. Per irRC criteria, Complete Response (irCR) is the disappearance of all target lesions, Partial Response (irPR) is a decrease in tumor burden by 50% or greater by a consecutive assessment at least 4 weeks after first documentation, Stable Disease (irSD) is the failure to meet criteria for irCR or irPR (in absence of irPD), Progressive Disease (irPD) is at least 25% increase in tumor burden relative to nadir. Estimation based on the Kaplan-Meier curve.
Time Frame: 28 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: MSI Positive Colorectal Cancer | Cohort B: MSI Negative Colorectal Cancer | Cohort C: MSI Positive Non-Colorectal Cancer
Number analyzed (Participants) | 41 | 25 | 47
percentage of participants | 70 [58 to 86] | 12 [4 to 36] | 64 [51 to 80]

8. Secondary Outcome: Objective Response Rate (ORR) in MSI Positive and Negative Solid Tumor Malignancies Using Response Evaluation Criteria in Solid Tumors (RECIST 1.1)
Description: ORR is defined as the percentage of patients achieving a complete response (CR) or partial response (PR) based on RECIST 1.1 criteria. CR = disappearance of all target lesions, PR is =>30% decrease in sum of diameters of target lesions.
Time Frame: 28 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: MSI Positive Colorectal Cancer | Cohort B: MSI Negative Colorectal Cancer | Cohort C: MSI Positive Non-Colorectal Cancer
Number analyzed (Participants) | 41 | 25 | 47
percentage of participants | 54 [37 to 69] | 0 [0 to 14] | 55 [40 to 70]

9. Secondary Outcome: Number of Patients Experiencing a Grade 3 or Above Treatment-related Toxicity
Description: When calculating the incidence of AEs, each adverse event (AE) (as defined by NCI CTCAE v4.03) will be counted only once for a given subject.
Time Frame: 28 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: MSI Positive Colorectal Cancer | Cohort B: MSI Negative Colorectal Cancer | Cohort C: MSI Positive Non-Colorectal Cancer
Number analyzed (Participants) | 41 | 25 | 47
Participants | 12 | 0 | 13

10. Secondary Outcome: Progression Free Survival (PFS) at 28 Weeks in MSI Positive and Negative Solid Tumor Malignancies Using Response Evaluation Criteria in Solid Tumors (RECIST 1.1)
Description: PFS is defined as the percentage of patients with disease progression (PD or relapse from CR as assessed using RECIST 1.1 criteria) or death due to any cause at 28 weeks. Per RECIST 1.1 criteria, CR = disappearance of all target lesions, Partial Response (PR) is =>30% decrease in sum of diameters of target lesions, Progressive Disease (PD) is >20% increase in sum of diameters of target lesions, Stable Disease (SD) is <30% decrease or <20% increase in sum of diameters of target lesions. Estimation based on the Kaplan-Meier curve.
Time Frame: 28 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: MSI Positive Colorectal Cancer | Cohort B: MSI Negative Colorectal Cancer | Cohort C: MSI Positive Non-Colorectal Cancer
Number analyzed (Participants) | 41 | 25 | 47
percentage of participants | 70 [57 to 86] | 16 [6 to 41] | 64 [51 to 79]

11. Secondary Outcome: Disease Control Rate in MSI Positive and Negative Solid Tumor Malignancies Using Response Evaluation Criteria in Solid Tumors (RECIST 1.1)
Description: Disease Control Rate (DCR) is defined as the percentage of patients achieving a complete response (CR) or partial response (PR) or stable disease (SD) based on RECIST 1.1 criteria. CR = disappearance of all target lesions, PR is =>30% decrease in sum of diameters of target lesions, progressive disease (PD) is >20% increase in sum of diameters of target lesions, stable disease (SD) is <30% decrease or <20% increase in sum of diameters of target lesions.
Time Frame: 28 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: MSI Positive Colorectal Cancer | Cohort B: MSI Negative Colorectal Cancer | Cohort C: MSI Positive Non-Colorectal Cancer
Number analyzed (Participants) | 41 | 25 | 47
percentage of participants | 80 [65 to 91] | 16 [5 to 36] | 70 [55 to 83]

12. Secondary Outcome: Does MSI as a Marker Predict Treatment Response
Description: ORR was used to determine whether MSI is a marker that predicts treatment response. This is the same data presented in outcome measure number 8 (ORR, to test against null of 5%).
Time Frame: 28 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: MSI Positive Colorectal Cancer | Cohort B: MSI Negative Colorectal Cancer | Cohort C: MSI Positive Non-Colorectal Cancer
Number analyzed (Participants) | 41 | 25 | 47
percentage of participants | 54 [37 to 69] | 0 [0 to 14] | 55 [40 to 70]

ADVERSE EVENTS:
Time Frame: 2 years 4 months Study treatment was administered for up to 2 years. Adverse events were accessed through 90 days after the last dose of study treatment.
Arm/Group | Cohort A: MSI Positive Colorectal Cancer | Cohort B: MSI Negative Colorectal Cancer | Cohort C: MSI Positive Non-Colorectal Cancer
All-Cause Mortality (participants affected / at risk) | 3/41 | 0/25 | 2/47
Serious Adverse Events (participants affected / at risk) | 4/41 | 0/25 | 7/47
Other Adverse Events (participants affected / at risk) | 41/41 | 3/25 | 47/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: MSI Positive Colorectal Cancer (N=41) | Cohort B: MSI Negative Colorectal Cancer (N=25) | Cohort C: MSI Positive Non-Colorectal Cancer (N=47)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Infusion reaction (Product Issues) | 1 (1) | 0 (0) | 0 (0)
Neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase Increased (ALT) (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (AST) (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Alkaline Phosphate elevated (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
hemolytic anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: MSI Positive Colorectal Cancer (N=41) | Cohort B: MSI Negative Colorectal Cancer (N=25) | Cohort C: MSI Positive Non-Colorectal Cancer (N=47)
Anemia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 4 (4)
Hypothyroidism/thyroiditis (Endocrine disorders) | 6 (6) | 0 (0) | 13 (13)
Diarrhea (Gastrointestinal disorders) | 10 (10) | 0 (0) | 9 (9)
Nausea (Gastrointestinal disorders) | 5 (5) | 0 (0) | 8 (8)
Fatigue (General disorders) | 8 (8) | 1 (1) | 13 (13) — and administration site conditions
Alanine aminotransferase Increased (ALT) (Investigations) | 3 (3) | 0 (0) | 3 (3)
Aspartate aminotransferase increased (AST) (Investigations) | 4 (4) | 0 (0) | 5 (5)
Lymphocyte count decreased (Investigations) | 2 (2) | 0 (0) | 5 (5)
White blood cell decreased (Investigations) | 3 (3) | 0 (0) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 0 (0) | 4 (4)
Neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 5 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (6) | 0 (0) | 13 (13)
Rash (Skin and subcutaneous tissue disorders) | 10 (10) | 2 (2) | 15 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-01): https://cdn.clinicaltrials.gov/large-docs/11/NCT01876511/Prot_SAP_000.pdf